CLINICAL TRIAL: NCT02933801
Title: ODM-201 Maintenance Therapy in Patients With Metastatic Castration Resistant Prostate Cancer (mCRPC) Previously Treated With Novel Hormonal Agents and Non-progressive Disease After Subsequent Treatment With a Taxane: A Multicenter Randomized Double-blind Placebo-controlled Phase II Trial.
Brief Title: ODM-201 Maintenance Therapy in Patients With mCRPC Previously Treated With Novel Hormonal Agents.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Decision Board no further financial support after 3 years of follow-up as remaining patients in follow-up phase would not relevantly change the endpoints.
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAKK 08/16; 2016-003996-23 (EudraCT Number)
Record Dates: First submitted 2016-10-13; First posted 2016-10-14 (Estimated); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Prostate Cancer Metastatic; Prostate Cancer
Keywords: metastatic castration resistant prostate cancer (mCRPC); Prostate Cancer; phase II trial; ODM-201; maintenance therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — darolutamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: ODM-201 (Experimental): 600mg ODM-201 BID (twice daily) and Best Supportive Care until progression
  Interventions: Drug: ODM-201
- Arm B: Placebo (Placebo Comparator): Placebo BID (twice daily) and Best Supportive Care until progression
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ODM-201 — ODM-201 will be given at a dose of 600 mg BID orally on a continuous basis.
  Other Names: BAY-1841788
  Arms: Arm A: ODM-201
Other: Placebo — Placebo will be given at a dose of 600 mg BID orally on a continuous basis.
  Arms: Arm B: Placebo

SUMMARY:
The main objective of the trial is to assess impact of maintenance therapy with ODM-201 on radiographic progression-free survival (rPFS) of patients with mCRPC pretreated with novel hormonal agents who have non-progressive disease after chemotherapy with a taxane.

DETAILED DESCRIPTION:
The treatment of metastatic castration-resistant prostate cancer has evolved rapidly over the past few years. First line treatment with one of the novel antihormonal drugs abiraterone or enzalutamide followed by chemotherapy with docetaxel is now standard of care. If a patient has disease stabilization on chemotherapy he undergoes a watchful waiting period and further treatment is only started at the time of disease progression. This trial tests the immediate use of the novel androgen receptor antagonist ODM-201 as maintenance treatment after chemotherapy aiming at prolonging radiographic progression free survival as compared to watchful waiting.

The main objective of the trial is to assess impact of maintenance therapy with ODM-201 on radiographic progression-free survival (rPFS) of patients with mCRPC pretreated with novel hormonal agents who have non-progressive disease after chemotherapy with a taxane.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to Swiss law and ICH/GCP regulations before registration and prior to any trial specific procedures not part of normal medical care.
* Histologically or cytologically confirmed diagnosis of adenocarcinoma of the prostate
* Castration resistance: tumor progression after orchiectomy or during treatment with GnRH analogues (agonists or antagonists)
* Metastatic disease, documented by imaging
* Total testosterone ≤ 50 ng/dL (≤ 1.7 nmol/L)
* Treatment with abiraterone AND/OR enzalutamide for at least 8 weeks prior to taxane based chemotherapy
* No evidence of disease progression after chemotherapy with docetaxel (at least cumulative dose of ≥ 300 mg/m2 or total dose ≥ 600mg) or cabazitaxel (at least cumulative dose of ≥ 80 mg/m2 or total dose ≥ 160 mg)

  * No evidence of progression on imaging according to PCWG3
  * No evidence of progression on PSA levels referred to the nadir since start of taxane treatment (PSA progression defined as > 25% increase of PSA level or >50% if PSA decrease under chemotherapy >50% AND > 5 ng/mL increase in the absolute PSA value)
* Non-surgically castrated patient agrees on ongoing use of GnRH analogues (agonists or antagonists) during the trial
* Planned start of trial treatment 2 to 8 weeks after last taxane dose
* Male patient 18 years or older
* WHO performance status of ≤2
* Laboratory values as specified below

  * alanine aminotransferase (ALT) ≤ 2.5 x ULN (except for patients with liver metastases ≤ 5.0 x ULN)
  * Total bilirubin ≤ 1.5 x ULN (except for patients with Gilbert's disease ≤ 3.0 x ULN)
  * Estimated creatinine clearance using the Cockcroft-Gault formula > 30 mL/minute
  * Blood counts at screening: haemoglobin ≥ 90 g/L, absolute neutrophil count ≥ 1500/μl (1.5x109/L), platelet count ≥ 100,000/μl (100x109/L) (patient must not have received any growth factor or blood transfusion within 7 days of the haematology laboratory obtained at screening)
* Adequate cardiac function: Left ventricular Ejection Fraction (LVEF) ≥ 40% as determined by echocardiography (ECHO)
* Patient is able and willing to swallow trial drug as whole tablet
* Sexually active male subjects must agree to use condoms as an effective barrier method and refrain from sperm donation, and/or their female partners of reproductive potential to use a method of effective birth control, during the study treatment and for 3 months after the end of the treatment.
* Patient agrees to participate in the mandatory translational research project

Exclusion Criteria:

* Prior chemotherapy for prostate cancer except from chemotherapy with a taxane
* Concurrent disease requiring higher doses of corticosteroid than the equivalent of 10 mg prednisone per day
* Known CNS or leptomeningeal metastases
* Clinical or radiological evidence of current spinal cord compression
* History of hematologic or primary solid tumor malignancy, unless in remission for at least 2 years from registration with the exception of localized non-melanoma skin cancer or carcinoma in situ having undergone complete resection.
* Prior therapy for mCRPC with modern anti-hormonal treatment except for enzalutamide or abiraterone
* Concurrent treatment with other experimental drugs or treatment in a clinical trial within 30 days prior to trial entry (except clinical trial SAKK 96/12)
* Concomitant use of other anti-cancer drugs or radiotherapy except for local pain control and GnRH analogues
* Severe or uncontrolled cardiovascular disease
* Acute exacerbations of chronic illnesses, serious infections, or major surgery within 4 weeks before expected start of treatment
* ECG abnormalities of Q-wave infarction, unless identified ≥ 6 months prior to registration or QTc interval >480 msec
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the GI absorption or tolerance of ODM-201
* Known hypersensitivity to trial drug or to any component of the trial drug
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Radiographic progression-free survival (rPFS) at 12 weeks | At 12 weeks after treatment start
  Radiographic progression-free survival is defined as the time from treatment start to radiographic disease progression or death from any cause, whichever occurs earlier.

SECONDARY OUTCOMES:
Radiographic progression-free survival (rPFS) | Every 12 weeks until disease progression (estimated up to 1 year)
  Radiographic progression-free survival is defined as the time from treatment start to radiographic disease progression or death from any cause, whichever occurs earlier.
Time to PSA progression | PSA level at baseline and every 4 weeks until disease progression (estimated up to 1 year)
  PSA progression is defined as:
  * In case PSA levels had not decreased under treatment with the study drug: ≥ 25% increase over baseline (last PSA measurement before treatment start) AND an increase in the absolute PSA value of ≥ 5 ng/mL.
  * In case of PSA response < 50% under treatment with the study drug: ≥ 25% increase over the nadir AND an increase in the absolute PSA value of ≥ 5 ng/mL.
  * In case of PSA response ≥ 50% under treatment with the study drug: ≥ 50% increase over the nadir AND an increase in the absolute PSA value of ≥ 5 ng/mL
Time to symptomatic/clinical progression | treatment start to the time point of symptomatic/clinical progression (estimated up to 1 year)
  Symptomatic/clinical progression is defined by one of the following:
  * Occurrence of a SRE due to bone metastases, defined as pathologic fracture, spinal cord compression, palliative radiation to bone, or surgery to bone
  * Treating physician decides for intervention due to new disease related complications (e.g., urinary obstruction, hydronephrosis)
Event-free survival | treatment start until the event of interest (estimated up to 1 year)
  Event-free survival is defined as the time from treatment start until the event of interest.
Overall survival | time from trial randomization to the date of death from any cause (estimated up to 6 years)
  Overall survival is defined as the time from treatment start until death from any cause.
PSA response (30%, 50%, 90% and best) | PSA level at baseline and every 4 weeks until disease progression (estimated up to 1 year)
  30% PSA response is defined as a decrease in PSA level of at least 30% (compared to baseline PSA).
  50% PSA response is defined as a decrease in PSA level of at least 50% (compared to baseline PSA).
  90% PSA response is defined as a decrease in PSA level of at least 90% (compared to baseline PSA).
  Best PSA response is defined as the percentage of change in PSA from baseline to the maximum decline in PSA at any point under treatment. If there is a steady increase after baseline, the best response is defined as the percentage of change in PSA from baseline to the minimum increase in PSA at any point under treatment. Baseline is defined as the latest recorded measurement prior to the first dose of trial treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Silke Gillessen, Prof, Study Chair — Cantonal Hospital of St. Gallen
Locations (32):
- France (4):
  - Institut Bergonié, Bordeaux
  - Centre Oscar Lambret, Lille
  - Centre de lutte contre le cancer Léon Bérard, Lyon
  - Centre Eugène Marquis, Rennes
- Italy (8):
  - European Institute of Oncology (EIO), Milan
  - Istituto Nazionale dei Tumori - IRCCS Fondazione, Milan
  - Istituto Nazionale dei Tumori - IRCCS Fondazione Pascale S.C., Napoli
  - AOU "Maggiore della Carità" di S.C. di Oncologia, Novara
  - AOU San Luigi Gonzaga, Orbassano
  - AO San Camillo and Forlanini Hospitals, Roma
  - Presidio Ospedaliero Santa Chiara, Trento
  - Azienda Ospedaliera Universitaria Integrate Verona (AOUI), Verona
- Spain (10):
  - Hospital de Torrecárdenas, Almería
  - Hospital Universitario Infanta Cristina, Badajoz
  - Hospital Clinic Barcelona, Barcelona
  - Consorcio Hospitalario Provincial de Castellon, Castellon
  - Hospital Universitario San Cecilio, Granada
  - Hospital Univ. de Guadalajara, Guadalajara
  - Centro Integral Oncológico Clara Campal - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario Puerta de Hierro-Majadahonda, Majadahonda
  - Hospital General Universitario Morales Meseguer, Murcia
  - Complejo Hospital Universitario de Santiago de Compostela, Santiago de Compostela
- Switzerland (10):
  - Kantonsspital Baden, Baden
  - Istituto Oncologico della Svizzera Italiana (IOSI), Bellinzona
  - Kantonsspital Graubuenden, Chur
  - Hôpital Fribourg HFR, Fribourg
  - Kantonsspital Liestal, Liestal
  - Fondazione Oncologia / Oncologia ematologia, Locarno
  - Kantonsspital Muensterlingen, Münsterlingen
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Hôpital du Valais (Sion et Martigny), Sion
  - Spital STS AG, Thun

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gillessen S, Procopio G, Hayoz S, Kremer E, Schwitter M, Caffo O, Lorente D, Pedrazzini A, Roubaud G, Nenan S, Omlin A, Buttigliero C, Delgado Mingorance JI, Gonzalez-Del-Alba A, Delgado MT, Nole F, Turco F, Pereira Mestre R, Ribi K, Cathomas R. Darolutamide Maintenance in Patients With Metastatic Castration-Resistant Prostate Cancer With Nonprogressive Disease After Taxane Treatment (SAKK 08/16). J Clin Oncol. 2023 Jul 10;41(20):3608-3615. doi: 10.1200/JCO.22.01726. Epub 2023 Feb 8. PMID 36753698